CLINICAL TRIAL: NCT04455724
Title: Negative Pressure Incisional Wound Therapy for High-risk Ventral Hernia Repair: a Randomized Controlled Trial
Brief Title: Negative Pressure Incisional Wound Therapy for High-risk Ventral Hernia Repair
Acronym: N-PITH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8183
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Given the physical differences in the negative pressure wound therapy systems compared to standard sterile dressings, patient participants and care providers will not be able to be blinded. Ultrasound evaluators and statisticians, however, will be.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Negative Pressure Incisional Wound Therapy (Experimental): A PREVENA™ PEEL & PLACE™ system kit will be applied to the surgical wound and assembled in the operating room following closure by primary intent. The system will be set for a negative pressure of -125mmHg. The dressing will be left in place for 7 days post-operation, during which the patient may be discharged from hospital. The dressing will only be removed or changed if the treating physician has suspicion of one of the complications included in the primary composite outcome or is planning re-intervention on the surgical site.
  Interventions: Device: Negative pressure incisional wound therapy
- Standard sterile dressing (Active Comparator): A sterile island dressing will be applied to the surgical wound in the operating room following closure by primary intent, which will be removed on post-operative day 2 and left open to air unless there is ongoing discharge.
  Interventions: Device: Standard sterile dressing

INTERVENTIONS:
Device: Negative pressure incisional wound therapy — A vacuum-style dressing system that is sealed in place over a surgical wound, applying constant negative pressure to the healing tissues.
  Arms: Negative Pressure Incisional Wound Therapy
Device: Standard sterile dressing — A standard, sterile island dressing
  Arms: Standard sterile dressing

SUMMARY:
The investigators are testing the ability of vacuum dressings to improve wound healing for patients having large hernias surgically repaired who are at risk of having wound complications. The trial will randomly be giving some patients having this surgery the vacuum dressing and some a standard dressing and observing how their wounds heal in hospital and at follow-up appointments.

DETAILED DESCRIPTION:
This study is a multicentre, clinical randomized controlled trial comparing the use of incisional negative pressure wound therapy versus standard sterile dressings in high-risk ventral hernia repairs. The trial will be enrolling patients undergoing elective or emergent ventral hernia repair who have risk factors for surgical wound complications and randomizing them to either receive a PREVENA incisional negative pressure wound therapy system dressing for 7 days post-operatively or a standard sterile dressing.for 2 days post-operatively. The primary outcome will be a composite of a variety of surgical site complications including wound infection, dehiscence, seroma / hematoma formation, non-healing wound, early hernia recurrence, and fistula formation. These will be evaluated by unblinded clinical judgement of treating physicians, and blinded assessment with ultrasonography. Secondary outcomes will include perceived difference in Quality of Life and cost-effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. patients undergoing surgical repair of ventral or incisional hernias greater than 3 cm in largest diameter
2. have one or more of the following risk factors for post-operative surgical site complications:

   1. Body Mass Index (BMI) greater than or equal to 30
   2. diagnosis of diabetes mellitus (either type I or II)
   3. previous history of hernia recurrence
   4. active smoker
   5. presence of colostomy or ileostomy
   6. age greater than 64
   7. chronic obstructive pulmonary disease
   8. chronic kidney disease
   9. clinically immunocompromised.

Exclusion Criteria:

1. the abdomen is left open post-operatively, or
2. if the patient has a sensitivity to silver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Surgical Site Complications | First 3 months post-operatively
  Composite of incidence of surgical site infection, hematoma formation, seroma formation, wound dehiscence, hernia recurrence, and fistula formation.

SECONDARY OUTCOMES:
Quality of life after surgery: survey | 3 months post-operatively
  Quality of life as measured using the Hernia-Related Quality of Life Survey (HerQLes). Scoring is out of 100, with higher scores indicating better quality of life.
Cost-effectiveness | 3 months post-operatively
  Cost in dollars per quality-adjusted life year, measured using hospital length of stay, cost of complications, and cost of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Christopher E Blewett, MD, Principal Investigator — McMaster University
Locations (1):
- Niagara Health St. Catharines Site, St. Catharines, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindmark M, Strigard K, Lowenmark T, Dahlstrand U, Gunnarsson U. Risk Factors for Surgical Complications in Ventral Hernia Repair. World J Surg. 2018 Nov;42(11):3528-3536. doi: 10.1007/s00268-018-4642-6. PMID 29700567
- [Background] Nguyen MT, Berger RL, Hicks SC, Davila JA, Li LT, Kao LS, Liang MK. Comparison of outcomes of synthetic mesh vs suture repair of elective primary ventral herniorrhaphy: a systematic review and meta-analysis. JAMA Surg. 2014 May;149(5):415-21. doi: 10.1001/jamasurg.2013.5014. PMID 24554114
- [Background] Lee L, Mata J, Landry T, Khwaja KA, Vassiliou MC, Fried GM, Feldman LS. A systematic review of synthetic and biologic materials for abdominal wall reinforcement in contaminated fields. Surg Endosc. 2014 Sep;28(9):2531-46. doi: 10.1007/s00464-014-3499-5. Epub 2014 Mar 12. PMID 24619334
- [Background] Castro PM, Rabelato JT, Monteiro GG, del Guerra GC, Mazzurana M, Alvarez GA. Laparoscopy versus laparotomy in the repair of ventral hernias: systematic review and meta-analysis. Arq Gastroenterol. 2014 Jul-Sep;51(3):205-11. doi: 10.1590/s0004-2803201400030008. PMID 25296080
- [Background] Fischer JP, Wink JD, Nelson JA, Kovach SJ 3rd. Among 1,706 cases of abdominal wall reconstruction, what factors influence the occurrence of major operative complications? Surgery. 2014 Feb;155(2):311-9. doi: 10.1016/j.surg.2013.08.014. PMID 24433774
- [Background] Lovecchio F, Farmer R, Souza J, Khavanin N, Dumanian GA, Kim JY. Risk factors for 30-day readmission in patients undergoing ventral hernia repair. Surgery. 2014 Apr;155(4):702-10. doi: 10.1016/j.surg.2013.12.021. Epub 2013 Dec 25. PMID 24612622
- [Background] Badia JM, Casey AL, Petrosillo N, Hudson PM, Mitchell SA, Crosby C. Impact of surgical site infection on healthcare costs and patient outcomes: a systematic review in six European countries. J Hosp Infect. 2017 May;96(1):1-15. doi: 10.1016/j.jhin.2017.03.004. Epub 2017 Mar 8. PMID 28410761
- [Background] Correa NF, de Brito MJ, de Carvalho Resende MM, Duarte MF, Santos FS, Salome GM, Ferreira LM. Impact of surgical wound dehiscence on health-related quality of life and mental health. J Wound Care. 2016 Oct 2;25(10):561-570. doi: 10.12968/jowc.2016.25.10.561. PMID 27681586
- [Background] Gheorghe A, Moran G, Duffy H, Roberts T, Pinkney T, Calvert M. Health Utility Values Associated with Surgical Site Infection: A Systematic Review. Value Health. 2015 Dec;18(8):1126-37. doi: 10.1016/j.jval.2015.08.004. Epub 2015 Sep 26. PMID 26686800
- [Background] Guest JF, Fuller GW, Vowden P. Costs and outcomes in evaluating management of unhealed surgical wounds in the community in clinical practice in the UK: a cohort study. BMJ Open. 2018 Dec 14;8(12):e022591. doi: 10.1136/bmjopen-2018-022591. PMID 30552253
- [Background] Argenta LC, Morykwas MJ. Vacuum-assisted closure: a new method for wound control and treatment: clinical experience. Ann Plast Surg. 1997 Jun;38(6):563-76; discussion 577. PMID 9188971
- [Background] Capobianco CM, Zgonis T. An overview of negative pressure wound therapy for the lower extremity. Clin Podiatr Med Surg. 2009 Oct;26(4):619-31. doi: 10.1016/j.cpm.2009.08.002. PMID 19778692
- [Background] Ma Z, Li Z, Shou K, Jian C, Li P, Niu Y, Qi B, Yu A. Negative pressure wound therapy: Regulating blood flow perfusion and microvessel maturation through microvascular pericytes. Int J Mol Med. 2017 Nov;40(5):1415-1425. doi: 10.3892/ijmm.2017.3131. Epub 2017 Sep 13. PMID 28901392
- [Background] Morykwas MJ, Argenta LC, Shelton-Brown EI, McGuirt W. Vacuum-assisted closure: a new method for wound control and treatment: animal studies and basic foundation. Ann Plast Surg. 1997 Jun;38(6):553-62. doi: 10.1097/00000637-199706000-00001. PMID 9188970
- [Background] Orgill DP, Manders EK, Sumpio BE, Lee RC, Attinger CE, Gurtner GC, Ehrlich HP. The mechanisms of action of vacuum assisted closure: more to learn. Surgery. 2009 Jul;146(1):40-51. doi: 10.1016/j.surg.2009.02.002. Epub 2009 Apr 19. No abstract available. PMID 19541009
- [Background] Scherer SS, Pietramaggiori G, Mathews JC, Prsa MJ, Huang S, Orgill DP. The mechanism of action of the vacuum-assisted closure device. Plast Reconstr Surg. 2008 Sep;122(3):786-797. doi: 10.1097/PRS.0b013e31818237ac. PMID 18766042
- [Background] Moues CM, Vos MC, van den Bemd GJ, Stijnen T, Hovius SE. Bacterial load in relation to vacuum-assisted closure wound therapy: a prospective randomized trial. Wound Repair Regen. 2004 Jan-Feb;12(1):11-7. doi: 10.1111/j.1067-1927.2004.12105.x. PMID 14974959
- [Background] Dohmen PM, Markou T, Ingemansson R, Rotering H, Hartman JM, van Valen R, Brunott M, Segers P. Use of incisional negative pressure wound therapy on closed median sternal incisions after cardiothoracic surgery: clinical evidence and consensus recommendations. Med Sci Monit. 2014 Oct 4;20:1814-25. doi: 10.12659/MSM.891169. PMID 25280449
- [Background] Rodriguez-Unda N, Soares KC, Azoury SC, Baltodano PA, Hicks CW, Burce KK, Cornell P, Cooney CM, Eckhauser FE. Negative-Pressure Wound Therapy in the Management of High-Grade Ventral Hernia Repairs. J Gastrointest Surg. 2015 Nov;19(11):2054-61. doi: 10.1007/s11605-015-2894-0. Epub 2015 Aug 4. PMID 26239514
- [Background] Conde-Green A, Chung TL, Holton LH 3rd, Hui-Chou HG, Zhu Y, Wang H, Zahiri H, Singh DP. Incisional negative-pressure wound therapy versus conventional dressings following abdominal wall reconstruction: a comparative study. Ann Plast Surg. 2013 Oct;71(4):394-7. doi: 10.1097/SAP.0b013e31824c9073. PMID 22868327
- [Background] Pauli EM, Krpata DM, Novitsky YW, Rosen MJ. Negative pressure therapy for high-risk abdominal wall reconstruction incisions. Surg Infect (Larchmt). 2013 Jun;14(3):270-4. doi: 10.1089/sur.2012.059. Epub 2013 Apr 16. PMID 23590852
- [Background] Swanson EW, Cheng HT, Susarla SM, Lough DM, Kumar AR. Does negative pressure wound therapy applied to closed incisions following ventral hernia repair prevent wound complications and hernia recurrence? A systematic review and meta-analysis. Plast Surg (Oakv). 2016 Summer;24(2):113-8. Epub 2016 May 27. PMID 27441196
- [Background] Abesamis GM, Chopra S, Vickery K, Deva AK. A Comparative Trial of Incisional Negative-Pressure Wound Therapy in Abdominoplasty. Plast Reconstr Surg Glob Open. 2019 May 16;7(5):e2141. doi: 10.1097/GOX.0000000000002141. eCollection 2019 May. PMID 31333924
- [Background] Hussamy DJ, Wortman AC, McIntire DD, Leveno KJ, Casey BM, Roberts SW. Closed Incision Negative Pressure Therapy in Morbidly Obese Women Undergoing Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2019 Oct;134(4):781-789. doi: 10.1097/AOG.0000000000003465. PMID 31503147
- [Background] Ren H, Li Y. Severe complications after negative pressure wound therapy in burned wounds: two case reports. Ther Clin Risk Manag. 2014 Jul 1;10:513-6. doi: 10.2147/TCRM.S66117. eCollection 2014. PMID 25061310
- [Background] Li Z, Yu A. Complications of negative pressure wound therapy: a mini review. Wound Repair Regen. 2014 Jul-Aug;22(4):457-61. doi: 10.1111/wrr.12190. PMID 24852446
- [Background] Webster J, Liu Z, Norman G, Dumville JC, Chiverton L, Scuffham P, Stankiewicz M, Chaboyer WP. Negative pressure wound therapy for surgical wounds healing by primary closure. Cochrane Database Syst Rev. 2019 Mar 26;3(3):CD009261. doi: 10.1002/14651858.CD009261.pub4. PMID 30912582
- [Background] Yu L, Kronen RJ, Simon LE, Stoll CRT, Colditz GA, Tuuli MG. Prophylactic negative-pressure wound therapy after cesarean is associated with reduced risk of surgical site infection: a systematic review and meta-analysis. Am J Obstet Gynecol. 2018 Feb;218(2):200-210.e1. doi: 10.1016/j.ajog.2017.09.017. Epub 2017 Sep 23. PMID 28951263
- [Background] Stannard JP, Volgas DA, McGwin G 3rd, Stewart RL, Obremskey W, Moore T, Anglen JO. Incisional negative pressure wound therapy after high-risk lower extremity fractures. J Orthop Trauma. 2012 Jan;26(1):37-42. doi: 10.1097/BOT.0b013e318216b1e5. PMID 21804414
- [Background] Pachowsky M, Gusinde J, Klein A, Lehrl S, Schulz-Drost S, Schlechtweg P, Pauser J, Gelse K, Brem MH. Negative pressure wound therapy to prevent seromas and treat surgical incisions after total hip arthroplasty. Int Orthop. 2012 Apr;36(4):719-22. doi: 10.1007/s00264-011-1321-8. Epub 2011 Jul 15. PMID 21761149
- [Background] Masden D, Goldstein J, Endara M, Xu K, Steinberg J, Attinger C. Negative pressure wound therapy for at-risk surgical closures in patients with multiple comorbidities: a prospective randomized controlled study. Ann Surg. 2012 Jun;255(6):1043-7. doi: 10.1097/SLA.0b013e3182501bae. PMID 22549748
- [Background] Grauhan O, Navasardyan A, Hofmann M, Muller P, Stein J, Hetzer R. Prevention of poststernotomy wound infections in obese patients by negative pressure wound therapy. J Thorac Cardiovasc Surg. 2013 May;145(5):1387-92. doi: 10.1016/j.jtcvs.2012.09.040. Epub 2012 Oct 27. PMID 23111014
- [Background] Grauhan O, Navasardyan A, Tutkun B, Hennig F, Muller P, Hummel M, Hetzer R. Effect of surgical incision management on wound infections in a poststernotomy patient population. Int Wound J. 2014 Jun;11 Suppl 1(Suppl 1):6-9. doi: 10.1111/iwj.12294. PMID 24851729